CLINICAL TRIAL: NCT01322516
Title: Outcomes of Pandemic Influenza in Pregnancy: an Observational Cohort Study
Brief Title: Outcomes of Pandemic Influenza in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dalhousie University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Shelly McNeil, Principal Investigator, Dalhousie University
Other Study IDs: 114231
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal swabs and serum
Oversight: Data Monitoring Committee: No

SUMMARY:
We propose to follow a cohort of pregnant and post-partum Canadian women through the fall and winter of 2009/2010 and the anticipated second and third waves of the current pandemic in order to better understand the incidence, complications and risk factors for severe disease due to H1N1 influenza in pregnant women, and to contribute data on the safety and effectiveness of antivirals and vaccines in this population.

The primary hypotheses to be tested are:

(i) pandemic influenza infection in the second and third trimester of pregnancy is associated with an increase in adverse fetal outcomes (fetal loss, stillbirth, neonatal mortality, significant neonatal morbidity, prematurity) (ii) close contact with young children (<2 yrs) at home or work is the most important risk factor for influenza in pregnant women (iii) higher scores on a scale of community infection prevention (a combination of self-reported hand hygiene adherence, avoidance of ill persons and avoidance of crowds) are protective against influenza (iv) receipt of seasonal influenza vaccine from 2007 to 2009 will increase the risk of illness due to influenza A(H1N1)v in the second and third waves of the pandemic.

(v) pandemic influenza vaccine is effective in preventing symptomatic influenza in pregnant women.

(vi) vaccination of pregnant women against a particular strain of influenza protects their infants against influenza infection in the first six months of life.

DETAILED DESCRIPTION:
Subjects will be consented to participate in the study. They will complete a web-based baseline questionnaire. Participants will be given a nasal swab kit with instructions for obtaining swabs. Baseline blood (10mls) will be drawn for influenza serology and for measurement of total IgG and IgG subtypes. An email will be sent to each participant within 24 hours of their enrolment to welcome them to the study.

Participants will be asked to complete a weekly diary using web-based data entry. An email will be sent to each participant every Monday during the study reminding the participant to complete their weekly diary and to report and submit a nasal swab if they have any symptoms of an acute respiratory illness. Reminder emails will be sent 48 hours later if the weekly form remains incomplete. Participants will be telephoned if forms remain incomplete for three weeks. Weekly emails will also be used to update participants about vaccine availability, current vaccine recommendations, and any changes in expert recommendations for pregnant women.

Once every four weeks additional questions will be asked on the weekly survey. If any participant develops symptoms compatible with an acute viral respiratory illness they will be asked to collect and submit a nasal swab as soon as possible after the onset of symptoms and to complete an illness starting the day of symptom onset and ending when all symptoms are either absent or mild, or for 3 days, whichever is longer. Subjects will be notified if results are positive for influenza along with the local Medical Officer of Health. Treatment for influenza will be discussed with each infected participant by a physician investigator.

Repeat serology and blood for total IgG and IgG subtype will be drawn at the time of delivery to the six week post partum. Women will notify the study when they are admitted for delivery or termination of pregnancy and will be interviewed either in person at the hospital, or over the telephone within 3 weeks of delivery. A chart review will be performed to identify any complications at delivery or termination, and to record neonatal outcomes. Post-partum, mothers will continue their own weekly and illness diaries and weekly diaries for their infants will be added.

Pregnant women requiring hospital admission for influenza in hospitals participating in surveillance for the Toronto Invasive Bacterial Diseases Network (TIBDN) and Serious Outcomes Surveillance (SOS) for the PHAC/CIHR Influenza Research Network (PCIRN), as well as pregnant women with influenza admitted to intensive care units as part of the Canadian Critical Care Clinical Trials Group Influenza Surveillance System (ICU-Flu) will be approached. Risk factor data from the baseline and weekly questionnaires will be collected retrospectively from these women. With consent, women will be followed to delivery/termination, and the same information collected regarding neonatal outcomes as was collected for other women in the cohort.

An email will be sent to all participating women requesting their consideration of three additional parts of the study:

1. A questionnaire of development (the 8 month Ages and Stages® Questionnaire; see attached) to be completed by the parent
2. An assessment with a physical examination at 7-9 months of age by a trained physician or a nurse practitioner
3. Permission for the study to contact parents in the future about further follow-up.

Mothers will also be asked to book an appointment for the 7-9 month assessment. Mothers who do not wish to have a pediatrician assessment will be asked over the telephone if they have any questions they wish to have answered about the study or the Ages and Stages® questionnaire, and if they consent to contact for future long term follow-up studies. If the child's score on the Ages and Stages® questionnaire raises a concern, mothers will be offered the chance to discuss this with a study physician, to have the results shared with her child's physician and/or to be referred to a pediatrician.

Participants may choose to withdraw from the study at any time. When they do so, they will be asked if the data and blood samples that have been provided can be kept and used for study purposes. If a patient withdraws and cannot be contacted data that has been obtained will be retained, and blood will be used for the immediate study purpose, but will not be used for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Participants must:

  1. be and pregnant, and, at the time of enrolment, not more than 30 weeks gestation.
  2. be greater than or equal to 16 years of age
  3. give written informed consent prior to entry
  4. be available for follow-up during the study period
  5. have convenient access to a computer with internet access
  6. know basic skills for use of the internet
  7. have the ability to complete questionnaires in either English or French

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 800 pregnant women followed through pregnancy during second and third waves of the 2009 influenza pandemic, and 2009/10 influenza season. Forty percent are high risk pregnancies: either for maternal influenza complications (eg. underlying asthma, gestational diabetes mellitus in prior pregnancies) or high risk for obstetrical complications (eg. prior premature birth, multiple pregnancies). Recruitment from Halifax, Quebec City, Toronto, Hamilton, Calgary, Edmonton, and Vancouver. Plan to enroll all women before the beginning of the second wave; however, enrolment of women <20 weeks pregnant will continue at each site until the second wave has peaked locally.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-09; Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Influenza A(H1N1)v infection: will be as diagnosed by polymerase chain reaction(PCR) from nasal or nasopharyngeal (NP) swabs, and/or seroconversion to influenza A(H1H1)v. | October 2009 to June 2010
  Primary analysis for risk factors for infection will consider only symptomatic infection, defined as acute respiratory illness/ influenza like illness (fever (at least one measured T>=38°C) and cough and one other local or systemic symptom compatible with influenza) during the pregnancy with seroconversion to A(H1N1)v not explained by vaccination. Seroconversion defined as a 4 fold increase in hemagglutination inhibition titer from 1st to 2nd serum sample.
  Symptoms compatible with influenza defined as fever, cough, coryza, generalized myalgias, sore throat, headache, severe fatigue.

SECONDARY OUTCOMES:
Adverse fetal/neonatal outcome. | October 2009-June 2010
  Fetal loss >12 weeks, stillbirth, neonatal mortality, significant neonatal morbidity, prematurity, or low birth weight, stillbirth, neonatal mortality, prematurity, live birth at less than 37 weeks gestational age, low birth weight, significant neonatal morbidity, severe congenital malformation, complicated influenza infection.

CONTACTS AND LOCATIONS:
Overall Officials: Shelly McNeil, MD FRCPC, Principal Investigator — Dalhousie University, Halifax, NS; Emmanuel Bujold, MD, Principal Investigator — Laval University, Montreal, Quebec; Allison McGeer, MD FRCPC, Principal Investigator — University of Toronto, Toronto, Ontario; Mark Loeb, MD, Principal Investigator — McMaster University, Hamiton, Ontario; Marie Louie, MD, Principal Investigator — University of Calgary, Calgary, Alberta; George Zahariadis, MD, Principal Investigator — University of Alberta, Edmonton, Alberta; Deborah Money, MDFRCSC, Principal Investigator — University of British Columbia, Vancouver, British Columbia; Rachel Rodin, MD, Principal Investigator — Public Health Agency of Canada, Ottawa, Ontario
Locations (8):
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - University of Edmonton, Edmonton, Alberta
  - British Columbia's Women's and Children's Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Public Health Agency of Canada, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Laval University, Montreal, Quebec